CLINICAL TRIAL: NCT07351812
Title: Evaluation of Two Treatment Modalities for Myogenous Temporomandibular Disorders: A Randomized Controlled Trial
Brief Title: Two Treatment Modalities for Myogenous Temporomandibular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0999_11/2024
Record Dates: First submitted 2025-12-20; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: TMD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilization appliance (Experimental): Maxillary and mandibular impressions will be taken using irreversible hydrocolloid and poured immediately with Type IV dental stone to obtain study casts. A maxillary stabilization appliance will be fabricated according to Okeson et al. using 2-mm hard thermoplastic sheets. The appliance will have a flat occlusal surface with buccal extensions, and its fit and retention will be verified. Participants will wear the appliance for 3 months. Surface electromyography of the temporalis and masseter muscles will be recorded at baseline and after 3 months to assess changes in muscle activity
  Interventions: Other: Stabilization Appliance
- Ear stent (Active Comparator): Participants will undergo ENT evaluation to exclude ear pathology and remove cerumen. Ear impressions will be taken using soft addition silicone injected with a 3.5-mm syringe and sent to a hearing-aid laboratory for fabrication. The stent will be hollowed longitudinally to prevent hearing impairment. Patients will be instructed to wear the stent full-time, removing it only during meals, showering, or swimming
  Interventions: Other: Ear Stent

INTERVENTIONS:
Other: Stabilization Appliance — Participants will receive a maxillary stabilization appliance fabricated from 2-mm hard thermoplastic material using diagnostic casts. The appliance fit will be verified, and patients will be instructed to wear it for 3 months.
  Arms: Stabilization appliance
Other: Ear Stent — Participants will undergo ENT evaluation prior to ear impression taking. Custom ear stents will be fabricated from soft addition silicone and hollowed to prevent hearing impairment.
  Arms: Ear stent

SUMMARY:
Temporomandibular disorder (TMD) is a common condition with multifactorial etiology, including trauma, emotional stress, parafunctional habits, and occlusal discrepancies. TMD may be classified as myogenous, involving the masticatory and cervical muscles, or arthrogenous, affecting the temporomandibular joint structures. Management approaches range from noninvasive to invasive methods. The intraoral stabilization appliance (SA) is a widely used noninvasive treatment, while the ear stent (ES) has recently been introduced for managing myogenous TMD.

Aim: This randomized clinical trial aims to compare the effectiveness of SA and ES in the management of myogenous TMD.

ELIGIBILITY:
Inclusion Criteria:

* Participants presenting with pain score grading at least 4 out of 10 on NRS.
* Participants with fully dentate type I occlusion.
* Patients experiencing no neurological disorders.

Exclusion Criteria:

* Patients with arthrogenous TMJ will be excluded by Magnetic Resonance Imagining (MRI)
* Patients who have clicking or crepitation.
* Previous history of TMD treatment.
* History of recent trauma.
* The presence of systemic diseases (i.e., rheumatoid arthritis, osteoarthritis myologic or arthrological disease).
* Vascular disease (migraine and hypertension).
* Participants with uncontrolled systemic disease (diabetes), hematologic or neurologic disorders or inflammatory diseases.
* Patients who: Underwent trigger point myofascial injection, intramuscular stimulation, or dry needling in the last six months or Underwent neck and/or shoulder surgery in the last year.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle activity | Baseline and 3 months
  surface electromyography will be used to assess the temporalis and masseter muscles. The electrodes detect the electrical potentials generated by muscle fibers when they contract. This electrical activity is amplified and recorded by an electromyograph machine
Change in mouth opening | Baseline and 3 months
  Measure the distance (in mm) between the incisal edge of the maxillary and mandibular central incisors

SECONDARY OUTCOMES:
Change in pain | Baseline and 3 months
  NRS will be measured from the patient mark from 0 to 10, where 0 representing no pain and 10 representing the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt